CLINICAL TRIAL: NCT03175510
Title: Reliabılıty,Validity Of The Turkish Version Of The Back Pain Function Scale
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, GÖKHAN MARAŞ, Research assistant, Gazi University
Other Study IDs: 2017-72
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-06

CONDITIONS: Low Back Pain
Keywords: validity, reliability, low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients group: Patients with low back pain (18-65 years)

SUMMARY:
This study, we performed the Turkish version validity and reliability of the Back Pain Function Scale.

DETAILED DESCRIPTION:
Low back pain is defined as the pain that can occur in the region between the lower border of the scapula and the hip, sometimes spreading to the lower extremities, which causes activity limitation and is one of the most common health problems in the society. Appropriate use of assessment questionnaires is one of the most important steps in the evaluation of the functional level of the patient and in deciding on an effective treatment protocol. The purpose of our study is to determine the Turkish version, validity and reliability of Back Pain Function Scale. 180 patients with chronic low back pain were included in the study. Test-retest and internal consistency analysis were conducted to determine the reliability of the questionnaire. Test-retest results were evaluated using the Intraclass Correlation Coefficient method. Intraclass Correlation Coefficient results vary between 0.857 and 0.951, and the total Intraclass Correlation Coefficient value is found to be 0.961. These results indicate that the test-retest responses have a high degree of correlation. For internal consistency analysis, the Cronbach Alpha score was fou nd to be 0.910, indicating that the survey has high internal consistency. The total score obtained from the Back Pain Function Scale was assessed using the Pearson correlation analysis with the total scores obtained from the Roland Morris Disability Scale , Oswestry Disability Scale. Pearson's correlation coefficient was -0.840 with Oswestry Disability Scale of Back Pain Function Scale, Pearson's correlation coefficient was -0.803 with Roland Morris Disability Scale. The results show that the Back Pain Function Scale correlates perfectly with the Oswestry Disability Scale and the Roland Morris Disability Scale. In conclusion, Turkish version of Bac Pain Function Scale is valid and reliable.

ELIGIBILITY:
Inclusion Criteria:

Having a low back pain Literate

Exclusion Criteria:

pregnant canser trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic back pain between the ages of 18-65
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Roland Morris disability questionnaire | 10 minute
  Roland Morris Disability Questionnaire, a widely used health status measure for low back pain. The RMDQ can be used in research or clinical practice.

SECONDARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | 10 minute
  The Oswestry Disability Index (ODI) has become one of the principal condition-specific outcome measures used in the management of spinal disorders

CONTACTS AND LOCATIONS:
Overall Officials: seyit citaker, Study Chair — gazi üniversity
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR